CLINICAL TRIAL: NCT07178613
Title: Assessment of the Dose Safety and Efficacy of Serine Combined With Fluorouracil Drugs
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-2025-19
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Advanced Colorectal Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serine + Fluoropyrimidine Group (Other)
  Interventions: Drug: Serine（Oral）; Drug: Fluoropyrimidine Drugs

INTERVENTIONS:
Drug: Serine（Oral） — This study evaluates the dose safety and efficacy of serine in combination with fluoropyrimidine-based therapies. Primary objective: To determine the safety of oral serine administration.
  Secondary objectives: 1. To assess the preliminary efficacy of serine in the study population. 2. To establish the recommended Phase 2 dose for oral serine.
Drug: Fluoropyrimidine Drugs — This study evaluates the dose safety and efficacy of serine in combination with fluoropyrimidine-based therapies. Primary objective: To determine the safety of oral serine administration.
  Secondary objectives: 1. To assess the preliminary efficacy of serine in the study population. 2. To establish the recommended Phase 2 dose for oral serine.

SUMMARY:
This study evaluates the dose safety and efficacy of serine in combination with fluoropyrimidine-based therapies. Primary objective: To determine the safety of oral serine administration.

Secondary objectives: 1. To assess the preliminary efficacy of serine in the study population. 2. To establish the recommended Phase 2 dose for oral serine.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years (inclusive), male or female;
2. Patients with advanced colorectal cancer confirmed by histopathological or cytological examination, eligible for standard first-line treatment with fluorouracil-containing regimens.
3. Patients must have at least one measurable lesion.
4. ECOG performance status ≤ 2.
5. Expected survival ≥ 3 months;
6. Major organ functions are essentially normal, with laboratory tests meeting the following criteria:

   Hematology (no transfusion of blood or blood products within 7 days prior to testing; no use of G-CSF or other hematopoietic growth factors for correction):

   Absolute neutrophil count ≥1.5×10⁹/L ; Platelets ≥75×10⁹/L ; Hemoglobin ≥90 g/L;

   Renal:

   Creatinine clearance (CrCl) or estimated glomerular filtration rate (eGFR) >60 mL/min/1.73 m² (Cockcroft-Gault formula);

   Liver:

   Serum total bilirubin <1.5×ULN; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5×ULN or ≤5×ULN (for subjects with liver metastases); Albumin (ALB) ≥30 g/L;

   Coagulation Function:

   International Normalized Ratio (INR) or Prothrombin Time (PT) < 1.5×ULN. If the subject is receiving anticoagulant therapy, PT is acceptable as long as it falls within the therapeutic range for the anticoagulant drug.

   Cardiovascular System:

   Ejection Fraction (EF) 55%-70%; QTc Interval: Male ≤440ms; Female ≤450ms.
7. Serum pregnancy tests for female subjects of childbearing potential during the screening period must be negative. Female/male subjects with reproductive potential must be willing to use reliable contraception throughout the study period (i.e., from signing the informed consent form until 90 days after the last study drug administration), including but not limited to: abstinence, male partner having undergone vasectomy, female sterilization, effective intrauterine device (IUD), and effective contraceptive medication.
8. Patients voluntarily participate in this study, sign informed consent forms, and demonstrate good compliance.

Exclusion Criteria:

1. Trial Participation Restrictions: Currently participating in or having received investigational drug/device treatment within the past 4 weeks;
2. Prior Fluorouracil-Based Therapy Restrictions: History of ≥Grade 3 toxicity (e.g., myelosuppression, gastrointestinal toxicity) following prior fluorouracil-based therapy, deemed unsuitable for re-administration by the investigator;
3. Recent Surgery Restriction: Undergone major surgery (excluding diagnostic biopsy) within 28 days prior to first dosing, or scheduled for surgery during the study period;
4. Metabolic and Nutritional Status Restriction: Presence of severe malnutrition (BMI < 18.5 or serum albumin < 30 g/L), or inability to supplement serine orally (e.g., malabsorption syndrome, short bowel syndrome); Known serine metabolism disorders (e.g., PHGDH/PSAT1 gene mutation-related diseases);
5. Concurrent severe disease restrictions: Severe cardiovascular disease (NYHA Class III/IV heart failure, myocardial infarction within 6 months, uncontrolled hypertension >150/100 mmHg); severe respiratory disease (COPD, GOLD Stage ≥3, interstitial lung disease); Active infection (requiring systemic antibiotic/antiviral therapy);
6. Active HIV/viral hepatitis: HIV-positive status, or active hepatitis B (HBV-DNA ≥ 2000 IU/mL), or active hepatitis C (HCV-RNA positive); (Note: Patients with HBV-DNA < 2000 IU/mL receiving antiviral therapy may be enrolled);
7. Neurological disorders: Uncontrolled brain metastases (with intracranial hypertension or neurological symptoms), or history of severe psychiatric illness/substance abuse (impeding treatment compliance);
8. Allergy history: Known allergy to fluorouracil-based drugs or serine supplements;
9. Pregnancy/lactation: Pregnant or lactating women (patients of childbearing potential must use highly effective contraception);
10. Other conditions deemed ineligible by the investigator: Any concomitant conditions or laboratory abnormalities that may interfere with study results, increase risk, or compromise patient safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety of Oral Serine | Up to 28 days
  Assess the safety of oral serine, including the occurrence of adverse events and dose - limiting toxicities